CLINICAL TRIAL: NCT00227760
Title: A Phase 2 Study of AZD2171 in Progressive Unresectable, Recurrent or Metastatic Renal Cell Carcinoma (RCC)
Brief Title: Cediranib Maleate in Treating Patients With Recurrent or Metastatic Kidney Cancer That Cannot Be Removed By Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2013-01072; NCI-2013-01072 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000446080; PHL-039 (Other: University Health Network Princess Margaret Cancer Center P2C); 7128 (Other: CTEP); N01CM62203 (NIH)
Record Dates: First submitted 2005-09-26; First posted 2005-09-28 (Estimated); Results first posted 2016-02-29 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2013-12

CONDITIONS: Recurrent Renal Cell Carcinoma; Stage IV Renal Cell Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — cediranib

ARMS (1):
- Treatment (cediranib maleate) (Experimental): Patients receive cediranib maleate PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cediranib Maleate; Procedure: Dynamic Contrast-Enhanced Magnetic Resonance Imaging; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study

INTERVENTIONS:
Drug: Cediranib Maleate — Given PO
  Other Names: AZD2171; AZD2171 Maleate; Recentin
Procedure: Dynamic Contrast-Enhanced Magnetic Resonance Imaging — Correlative studies
  Other Names: DCE MRI; DCE-MRI; DYNAMIC CONTRAST ENHANCED MRI
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase II trial studies how well cediranib maleate works in treating patients with recurrent or metastatic kidney cancer that cannot be removed by surgery. Cediranib maleate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the clinical benefit rate (objective response rate and rate of stable disease for at least 4 months) of AZD2171 (cediranib maleate) given to patients with progressive unresectable or, recurrent or metastatic renal cell carcinoma (RCC).

II. To assess the duration of response or stable disease, progression free, median and overall survival rates, and safety and tolerability of AZD2171.

III. To measure baseline and post treatment levels of soluble markers of angiogenic growth factors and receptors as well as levels of circulating endothelial cells, and correlate these with clinical outcome.

IV. To assess changes in blood flow and vessel permeability using dynamic contrast enhanced magnetic resonance imaging (DCE-MRI) pre and post treatment and to correlate these changes with clinical outcome.

OUTLINE:

Patients receive cediranib maleate orally (PO) once daily (QD) on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 4 weeks and then every 3 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed renal cell cancer that is locally recurrent or metastatic and is not considered curable by standard therapy
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as > 20 mm with conventional techniques or as > 10 mm with spiral computed tomography (CT) scan; bone lesions are not considered to be measurable; all radiology must be performed within 28 days prior to registration
* Previous therapy:

  * Surgery: Previous surgery is permissible; patients must be >= 4 weeks since any major surgery
  * Chemotherapy: No previous systemic chemotherapy
  * Immunotherapy: No previous therapy permitted
  * Gene/investigational therapy: No prior therapy is permitted
  * Radiation: Patients may have had radiation therapy but must have recovered from acute toxic effects prior to registration; at least 4 weeks must have elapsed since last dose of radiation before registration (exceptions may be made for low-dose, non-myelosuppressive radiotherapy); if the sole site of measurable disease is in a radiation field, there must have been documented progression at that site for patient to be eligible
* Life expectancy of greater than 3 months
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Absolute neutrophil count >= 1.5 x10^9/L
* Platelets >= 100 x10^9/L
* Total bilirubin =< 1.5 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 × institutional ULN
* Creatinine =< 1.5 x ULN OR creatinine clearance >= 60 mL/min/1.73 m^2
* AZD2171 has been shown to terminate fetal development in the rat, as expected for a process dependent on vascular endothelial growth factor (VEGF) signaling; for this reason, women of child-bearing potential must have a negative pregnancy test prior to study entry; women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had radiotherapy, or major surgery within 4 weeks prior to entering the study or those who have not recovered from adverse events of these therapies
* Patients may not be receiving any other investigational agents nor have participated in an investigational trial
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to AZD2171
* Mean corrected QT interval (QTc) > 470 msec (with Bazett's correction) in screening electrocardiogram or history of familial long QT syndrome
* Greater than +1 proteinuria on two consecutive dipsticks taken no less than 1 week apart
* Uncontrolled intercurrent illness including, but not limited to hypertension, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because AZD2171 is a VEGF inhibitor with known abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with AZD2171, breastfeeding should be discontinued if the mother is treated with AZD2171
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with AZD2171; appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated
* Any significant abnormality noted in the electrocardiogram (ECG) within 14 days of treatment
* A New York Heart Association classification of III or IV (NOTE: Patients classified as class II controlled with treatment may continue with increase monitoring)
* Conditions requiring concurrent use of drugs or biologics with proarrhythmic potential; these drugs are prohibited during studies with AZD2171

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2005-12; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Srikala Sridhar, Principal Investigator — University Health Network Princess Margaret Cancer Center P2C
Locations (6):
- Canada (6):
  - Cross Cancer Institute, Edmonton, Alberta
  - BCCA-Vancouver Cancer Centre, Vancouver, British Columbia
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - London Regional Cancer Program, London, Ontario
  - The Ottawa Hospital Cancer Centre (Ottawa Health Research Institute) Civic Campus, Ottawa, Ontario
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Cediranib Maleate)
Started | 44
Completed | 44
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Cediranib Maleate)
Number analyzed (Participants) | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 14
Age, Continuous [Median (Full Range); unit: years] | 62 [44 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 35
Region of Enrollment [Number; unit: participants]
  Canada | 44

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Durable Stable Disease, Evaluated Using the Response Evaluation Criteria in Solid Tumors (RECIST)
Description: Stable disease for a clinical benefit rate, evaluated using the Response Evaluation Criteria in Solid Tumors (RECIST)
Time Frame: 4 weeks
Population: Evaluable patients
Measure: Number; unit: particip[ants
Arm/Group | Treatment (Cediranib Maleate)
Number analyzed (Participants) | 39
particip[ants | 18

2. Primary Outcome: Objective Response, Evaluated Using RECIST
Description: Partial response as assessed by RECIST criteria
Time Frame: 4 weeks
Population: Evaluable patients
Measure: Number; unit: participants
Arm/Group | Treatment (Cediranib Maleate)
Number analyzed (Participants) | 39
participants | 15

3. Secondary Outcome: Progression Free Survival
Time Frame: Time from start of treatment to progression, death or last contact, or last tumor assessment before the start of further antitumor therapy, assessed up to 6.5 years
Population: Total patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Cediranib Maleate)
Number analyzed (Participants) | 44
months | 8.9 [5.1 to 12.9]

ADVERSE EVENTS:
Arm/Group | Treatment (Cediranib Maleate)
Serious Adverse Events (participants affected / at risk) | 21/44
Other Adverse Events (participants affected / at risk) | 2/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Cediranib Maleate) (N=44)
Thromboembolic event (Vascular disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 2 (2)
Syncope (Nervous system disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vascular disorder - other (Vascular disorders) | 1 (1)
Headache (Vascular disorders) | 3 (3)
Chest pain - cardiac (Cardiac disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Cediranib Maleate) (N=44)
Infection and infestations - other (Infections and infestations) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less